CLINICAL TRIAL: NCT04040088
Title: Utility of Gallium-68-DOTA-Octreotate PET/CT in the Characterization of Pediatric Neuroendocrine Tumors
Brief Title: An Investigational Scan (68Ga-DOTATATE PET/CT) in Diagnosing Pediatric Metastatic Neuroendocrine Tumors
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MC1872; NCI-2019-04392 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1872 (Other: Mayo Clinic in Rochester); 16-010137 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2019-07-19; First posted 2019-07-31 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Ganglioneuroblastoma; Ganglioneuroma; Neuroblastoma
MeSH Terms: conditions — Ganglioneuroblastoma; Ganglioneuroma; Neuroblastoma | interventions — Ga(III)-DOTATOC; gallium Ga 68 dotatate; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (68Ga-DOTATATE, PET/CT) (Experimental): Patients with newly diagnosed high-risk neuroendocrine cancer receive 68Ga-DOTATATE intravenously (IV) and undergo PET/CT over 20-30 minutes at diagnosis (before any treatment) and at the time of radiation treatment planning.
  Interventions: Procedure: Computed Tomography; Drug: Gallium Ga 68-DOTATATE; Procedure: Positron Emission Tomography
- Cohort B (68Ga-DOTATATE, PET/CT) (Experimental): Patients with previously diagnosed high-risk neuroendocrine cancer receive 68Ga-DOTATATE IV and undergo PET/CT over 20-30 minutes at the time of radiation treatment planning.
  Interventions: Procedure: Computed Tomography; Drug: Gallium Ga 68-DOTATATE; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Gallium Ga 68-DOTATATE — Given IV
  Other Names: (68)Ga-DOTA-TATE; 68Ga-DOTA-0-Tyr3-Octreotate; 68Ga-DOTATATE; Gallium Ga 68 Oxodotreotide; Gallium Oxodotreotide Ga-68; Gallium-68 DOTA-DPhe1, Tyr3-octreotate
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This trial studies how well an investigational scan called 68Ga-DOTATATE PET/CT works in diagnosing pediatric patients with neuroendocrine tumors that have spread to other places in the body (metastatic). A neuroendocrine tumor is an abnormal growth of neuroendocrine cells, which are cells resembling nerve cells and hormone-producing cells. 68Ga-DOTATATE is a radioactive substance called a radiotracer that when used with PET/CT scans, may work better than standard of care MIBG scans in diagnosing pediatric metastatic neuroendocrine tumors and targeting them with radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the difference in radiation therapy (RT) target volume definition between gallium Ga 68-DOTATATE (68Ga-DOTATATE) PET/CT and iobenguane (metaiodobenzylguanidine [MIBG]).

SECONDARY OBJECTIVES:

I. To estimate the difference in metastatic tumor burden as detected by 68Ga-DOTATATE PET/CT and MIBG.

II. To estimate the difference in metabolic activity between tumors diagnosed on 68Ga-DOTATATE PET/CT and MIBG.

III. To evaluate patterns of failure after RT in association with 68Ga-DOTATATE PET/CT and MIBG.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT A: Patients with newly diagnosed high-risk neuroendocrine cancer receive 68Ga-DOTATATE intravenously (IV) and undergo PET/CT over 20-30 minutes at diagnosis (before any treatment) and at the time of radiation treatment planning.

COHORT B: Patients with previously diagnosed high-risk neuroendocrine cancer receive 68Ga-DOTATATE IV and undergo PET/CT over 20-30 minutes at the time of radiation treatment planning.

After completion of study, patients are followed up per standard of care for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age =< 30 years
* Histological confirmation of neuroblastoma, ganglioneuroblastoma, or ganglioneuroma.
* High-risk neuroblastoma requiring consolidative RT, as determined by the treating radiation oncologist.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-3 (patients 16 years old or older at entry) or Lansky Score of 30-100 (patients <16 years old at entry).
* Planned for radiation planning and RT at enrolling institution.
* Documented negative pregnancy test prior to induction chemotherapy, for women of childbearing age within =< 7 days prior to registration.
* Willing to return to enrolling institution for follow-up imaging and clinical evaluation, or willing to send follow-up imaging and clinical notes to enrolling institution (during the observation phase of the study).

Exclusion Criteria:

* Pregnant women, nursing women who refuse to stop breastfeeding, or men/women of childbearing age who are unwilling to use an effective birth control method.
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Immunocompromised patients and patients known to be human immunodeficiency virus positive and currently receiving antiretroviral therapy. NOTE: Patients known to be human immunodeficiency virus positive, but without clinical evidence of an immunocompromised state, are eligible for this trial.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Difference in radiation treatment target volume definition between 68Ga-DOTATATE positron emission tomography/computed tomography (PET/CT) and iobenguane (MIBG) | From baseline to the time of radiation treatment planning (up to 3 months)
  Will analyze the data descriptively in lieu of hypothesis testing. However, each metastatic lesion will be analyzed independently. Will report the mean and standard deviation of the difference between target tumor volumes. For patients with more than one metastasis, will compute the difference in the sum of the target volumes for all metastases.

SECONDARY OUTCOMES:
Proportion of agreement between MIBG and 68Ga-DOTATATE PET/CT in identifying neuroendocrine tumors | At diagnosis and during the radiation treatment (RT) planning period (up to 3 months)
  Will calculate the proportion of metastatic tumors detected by MIBG that are also detected by 68Ga-DOTATATE PET/CT. Each metastatic lesion will be considered an independent data point. A 95% confidence interval will be included using the Clopper-Pearson method.
Tumor metabolic activity of 68Ga-DOTATATE PET/CT compared to MIBG | At diagnosis and during the RT planning period (up to 3 months)
  Will perform some descriptive analyses to note the differences between MIBG and 68Ga-DOTATATE PET/CT. This may include measuring the difference in the number of metastatic sites per patient. Each metastatic lesion will be considered an independent data point.
Patterns of failure after RT | Up to 2 years
  Will evaluate patterns of failure after RT and associate with MIBG and 68Ga-DOTATATE PET/CT using two-year relapse rates. Relapse is defined as an increase in treated lesion(s) and/or new tumor per the progressive disease category of the International Neuroblastoma Response Criteria. Two-year cumulative incidence of relapse from first day of RT for the four categories listed above will be calculated considering death as a competing risk. Each relapse site will be considered an independent event.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Laack, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials